CLINICAL TRIAL: NCT01335139
Title: A Randomized, Double-blind, Single-center, Placebo Controlled Study of Sublingual Immunotherapy and Subcutaneous Immunotherapy in Adults With Seasonal Allergic Rhinitis (ITN043AD)
Brief Title: Long-Term Effects of Sublingual Grass Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN043AD; 2010-023536-16 (EudraCT Number)
Record Dates: First submitted 2011-04-08; First posted 2011-04-14 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: sublingual immunotherapy; subcutaneous immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Sublingual Immunotherapy; Grazax

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SCIT + Placebo (Experimental): Subcutaneous immunotherapy (SCIT) + sublingual immunotherapy (SLIT) placebo
  Interventions: Biological: Subcutaneous immunotherapy (SCIT); Other: Placebo
- SLIT + Placebo (Experimental): Sublingual immunotherapy (SLIT) + subcutaneous immunotherapy (SCIT) placebo
  Interventions: Biological: Sublingual immunotherapy (SLIT); Other: Placebo
- Placebo + Placebo (Placebo Comparator): Sublingual immunotherapy (SLIT) placebo + subcutaneous immunotherapy (SCIT) placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Sublingual immunotherapy (SLIT) — Participants randomized to receive sublingual allergen tablet immunotherapy with placebo injections.
  Other Names: Grazax®
  Arms: SLIT + Placebo
Biological: Subcutaneous immunotherapy (SCIT) — Participants randomized to receive subcutaneous injection immunotherapy with placebo tablets. Subcutaneous immunotherapy was included as a positive control.
  Other Names: Alutard SQ Grass Pollen®
  Arms: SCIT + Placebo
Other: Placebo — Participants randomized to double-placebo tablets and injections. This group was included as a negative control.

SUMMARY:
The purpose of this research study is to investigate whether sublingual immunotherapy (SLIT, grass pollen tablets under the tongue) has long term effects in severe hay fever.

DETAILED DESCRIPTION:
This is a randomized, double-blind, single-center, placebo-controlled, three-arm study comparing SLIT with placebo and SCIT with placebo. The main comparison will be between SLIT and placebo.

Individuals with severe grass pollen hay fever, with or without associated seasonal asthma, will be recruited during the pollen season of March through September 2011. Eligible participants will be randomized to one of the following three treatment arms administered in a double-blind (masked), double-dummy fashion in a 1:1:1 ratio:

* SLIT + SCIT placebo
* SCIT + SLIT placebo
* SLIT placebo + SCIT placebo

Participants will receive treatment over a 2-year period followed by a 1-year blinded (masked) withdrawal phase. Participants will be provided with anti-allergic rescue medications (antihistamine, topical intranasal corticosteroids, and short-acting beta agonists) throughout the study. Clinical endpoint assessments will be performed at prior to initiating their assigned treatment, after 1 and 2 years of treatment, and after the 1-year withdrawal period at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* A clinical history of grass pollen-induced allergic rhinoconjunctivitis for at least 2 years with peak symptoms in May, June, or July;
* A clinical history of moderate to severe rhinoconjunctivitis symptoms interfering with usual daily activities or with sleep as defined according to the Allergic Rhinitis and its Impact on Asthma (ARIA) classification of rhinitis;
* A clinical history of rhinoconjunctivitis for at least 2 years requiring treatment with either antihistamines or nasal corticosteroids during the grass pollen season;
* Positive skin prick test response, defined as wheal diameter greater than or equal to 3 mm, to Phleum pratense (e.g., Timothy grass);
* Positive specific IgE, defined as greater than or equal to IgE class 2 (0.7 kU/L), against Phleum pratense;
* A positive response to nasal allergen challenge with Phleum pretense, defined as an increase in TNSS greater than or equal to 7 points above baseline;
* For women of childbearing age, a willingness to use an effective form of contraception for the duration of the trial; and
* The ability to give informed consent and comply with study procedures.

Exclusion Criteria:

* Prebronchodilator forced expiratory volume at 1 second (FEV1) less than 70% of predicted value at either screening or baseline visit;
* A clinical history of moderate to severe allergic rhinitis, according to the ARIA classification, due to tree pollen near or overlapping the grass pollen season;
* A clinical history of persistent asthma and/or requiring regular inhaled corticosteroids for > 4 weeks per year outside of the grass pollen season;
* A clinical history of moderate- severe allergic rhinitis, according to the ARIA classification, caused by an allergen to which the participant is regularly exposed;
* History of emergency visit or hospital admission for asthma in the previous 12 months;
* History of chronic obstructive pulmonary disease;
* History of significant recurrent acute sinusitis, defined as 2 episodes per year for the last 2 years, all of which required antibiotic treatment;
* History of chronic sinusitis, defined as a sinus symptoms lasting greater than 12 weeks that includes 2 or more major factors or 1 major factor and 2 minor factors. Major factors are defined as facial pain or pressure, nasal obstruction or blockage, nasal discharge or purulence or discolored postnasal discharge, purulence in nasal cavity, or impaired or loss of smell. Minor factors are defined as headache, fever, halitosis, fatigue, dental pain, cough, and ear pain, pressure, or fullness.
* At randomization, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media, or other relevant infectious process; serous otitis media is not an exclusion criterion. Participants may be re-evaluated for eligibility after symptoms resolve.
* Any tobacco smoking within the last 6 months or a history of ≥ 10 pack years;
* Previous treatment by immunotherapy with grass pollen allergen within the previous 5 years.
* Any history of grade 4 anaphylaxis due to any cause as defined by the World Allergy Organization (WAO) grading criteria for immunotherapy;
* History of bleeding disorders or treatment with anticoagulation therapy;
* History of anti-IgE monoclonal antibody treatment;
* Ongoing systemic immunosuppressive treatment;
* History of intolerance to the study therapy, rescue medications, or their excipients;
* For women of childbearing age a positive serum or urine pregnancy test with sensitivity of less than 50 mIU/mL within 72 hours before the start of study therapy;
* The use of any investigational drug within 30 days of the screening visit; or
* The presence of any medical condition that the investigator deems incompatible with participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Nasal Response to Allergen Challenge | 3 years
  Defined as the average of the Total Nasal Symptom Score (TNSS) area under the curve (AUC) measured at 0 to 1 hours and the AUC measured at 1 to 10 hours after allergen challenge. The primary outcome consists of the comparison of SLIT + SCIT placebo versus SLIT placebo + SCIT placebo.

SECONDARY OUTCOMES:
Skin Late Phase Response (LPR) to Intradermal Testing | Baseline (Time 0) and 1,-2, and -3 years
  Recorded as the mean diameter of the swelling measured at the specified time points after allergen challenge at 1, 2, and 3 years. The analysis of this outcome will compare the mean diameter of the swelling at 1, 2, and 3 years separately, adjusting for baseline diameter using ANCOVA at the 0.05 level of significance.
Skin Early Phase Response (EPR) to Intradermal Testing | Baseline (Time 0) and 1, -2, and -3 years
  Recorded as the mean diameter of the swelling measured at the specified time points after allergen challenge at 1, 2, and 3 years. The analysis of this outcome will compare the mean diameter of the swelling at 1, 2, and 3 years separately, adjusting for baseline diameter using ANCOVA at the 0.05 level of significance.
Nasal LPR | Baseline (Time 0) and 1, -2, and -3 years
  Defined as the TNSS AUC over the specified time periods after allergen challenge at 1, 2, and 3 years. The analysis of these this outcome will compare the mean TNSS AUC at 1, 2, and 3 years separately, adjusting for baseline LPR using ANCOVA at the 0.05 level of significance.
Nasal EPR | Baseline (Time 0) and 1, -2, and -3 years
  Defined as the TNSS AUC over the specified time periods after allergen challenge at 1, 2, and 3 years. The analysis of these this outcome will compare the mean TNSS AUC at 1, 2, and 3 years separately, adjusting for baseline EPR using ANCOVA at the 0.05 level of significance.
Peak Total Nasal Symptom Score (TNSS) EPR | Baseline (Time 0) and 1, -2, and -3 years
  Maximum TNSS score measured between 0 and 1 hour after challenge.
Peak Nasal Inspiratory Flow (PNIF) LPR | Baseline (Time 0) and 1, -2, and -3 years
  Defined as PNIF AUC over the specified time periods after allergen challenge at 1, 2 and 3 years. The analyses for this outcome will compare the mean PNIF AUC at 1, 2, and 3 years separately, adjusting for baseline PNIF using ANCOVA at the 0.05 level of significance.
Peak Nasal Inspiratory Flow (PNIF) LPR Area Under the Curve (AUC) | Baseline (Time 0) and 1, -2, and -3 years
  Defined as PNIF AUC over the specified time periods after allergen challenge at 1, 2 and 3 years. The analyses for this outcome will compare the mean PNIF AUC at 1, 2, and 3 years separately, adjusting for baseline PNIF using ANCOVA at the 0.05 level of significance.
Peak Nasal Inspiratory Flow (PNIF) EPR Area Under the Curve (AUC) | Baseline (Time 0) and 1, -2, and -3 years
  Defined as PNIF AUC over the specified time periods after allergen challenge at 1, 2 and 3 years. The analyses for this outcome will compare the mean PNIF AUC at 1, 2, and 3 years separately, adjusting for baseline PNIF using ANCOVA at the 0.05 level of significance. AUC measured hourly between 1 and 10 hours after challenge.
Skin Prick Test Endpoint Titration | Baseline (Time 0) and 1, -2, and -3 years
  Assessed as the mean wheal diameters (mm) in response to skin prick tests in duplicate with 1000 SQ, 10,000 SQ and 100,000 SQ units of grass pollen allergen.
Use of Rescue Medications During the Pollen Season | 1, -2, and -3 years
  A composite rescue medication score will be derived using a pre-defined scoring algorithm.
Mini Rhinoconjunctivitis Quality-of-Life Questionnaire Score | 1, -2, and -3 years
  Mini Rhinoconjunctivitis Quality-of-Life Questionnaire (MiniRQLQ) scores will be collected pre-, peak-, and post-pollen season at 1, 2, and 3 years.
Hay Fever Severity Score | 1, 2 and 3 years
  Measured at the end of each pollen season at 1, -2, and -3 years.
Weekly Visual Analog Symptom (VAS) Scores | 1, -2, and -3 years
  Weekly Visual Analogue Scale scores will be summarized descriptively by group and year.
EXPLORATORY: Mechanistic Assessments of Local Immune Responses | 1, 2, and 3 years
  Measured in the nasal mucosa before and after nasal allergen challenge. Nasal secretions will be assayed for inflammatory mediators and local antibodies.
EXPLORATORY: Mechanistic Assessments of Peripheral Blood Subsets | 1, 2, and 3 years
  Peripheral blood mononuclear cells (PBMCs) samples will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Durham, MD, Study Chair — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal. ITN TrialShare makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Background] Cox LS. Sublingual Immunotherapy for Allergic Rhinitis: Is 2-Year Treatment Sufficient for Long-term Benefit? JAMA. 2017 Feb 14;317(6):591-593. doi: 10.1001/jama.2017.0128. No abstract available. PMID 28196239
- [Result] Scadding GW, Calderon MA, Shamji MH, Eifan AO, Penagos M, Dumitru F, Sever ML, Bahnson HT, Lawson K, Harris KM, Plough AG, Panza JL, Qin T, Lim N, Tchao NK, Togias A, Durham SR; Immune Tolerance Network GRASS Study Team. Effect of 2 Years of Treatment With Sublingual Grass Pollen Immunotherapy on Nasal Response to Allergen Challenge at 3 Years Among Patients With Moderate to Severe Seasonal Allergic Rhinitis: The GRASS Randomized Clinical Trial. JAMA. 2017 Feb 14;317(6):615-625. doi: 10.1001/jama.2016.21040. PMID 28196255
- [Derived] Altman MC, Segnitz RM, Larson D, Jayavelu ND, Smith MT, Patel S, Scadding GW, Qin T, Sanda S, Steveling E, Eifan AO, Penagos M, Jacobson MR, Parkin RV, Shamji MH, Togias A, Durham SR. Nasal and blood transcriptomic pathways underpinning the clinical response to grass pollen immunotherapy. J Allergy Clin Immunol. 2023 Nov;152(5):1247-1260. doi: 10.1016/j.jaci.2023.06.025. Epub 2023 Jul 15. PMID 37460024
- See also: National Institute of Allergy and Infectious Disease (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org/
- See also: Immune Tolerance Network (ITN) TrialShare: open public access to participant-level data available for this trial — http://www.itntrialshare.org
- See also: University of California, San Francisco (UCSF) — http://www.ucsf.edu/
- See also: Imperial College London — http://www3.imperial.ac.uk/
- Available data/document: Individual Participant Data Set: ITN043AD — https://www.itntrialshare.org/project/Studies/ITN043ADJAMA/Study%20Data/begin.view — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.Creating an account for ITN TrialShare is free and allows for searching studies of interest.
- Available data/document: Synopsis, Adverse Events, -Data and Reports, -Schedule of Assessments: ITN043AD — https://www.itntrialshare.org/project/Studies/ITN043ADJAMA/Study%20Data/begin.view — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.Creating an account for ITN TrialShare is free and allows for searching studies of interest.